CLINICAL TRIAL: NCT02813512
Title: Adipose-Derived Stem Cells (ADSCs) Injections for Stroke
Brief Title: Clinical Trial Study About Human Adipose-Derived Stem Cells in the Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gwo Xi Stem Cell Applied Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH102-REC1-034
Record Dates: First submitted 2016-06-03; First posted 2016-06-27 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GXNPC1 (Experimental): Three subjects will be to treatment (n=3) groups. The treatment group will receive brain transplants of autologous ADSCs. Treatment group will receive rehabilitation after the transplantation. Subjects will be assessed by magnetic resonance imaging (MRI) and four standardized stroke indices: National Institutes of Health Stroke Scale (NIHSS), European Stroke Scale (ESS), European Stroke Motor Subscale (EMS), Barthel Index, MMSE and Gait analyses at 1 month, 3 months, and 6 months after treatment.
  Interventions: Drug: ADSCs

INTERVENTIONS:
Drug: ADSCs — Autologous ADSCs
  Other Names: hADSCs

SUMMARY:
The objective of the study is to confirm the safety and possible efficacy of Adipose-Tissue Derived Stem Cells treatment of chronic stroke. Specifically, the study will transplant autologous ADSCs into brain surrounding ischemic infarct in adult (65-80 years old) subjects who have chronic non-hemorrhagic stroke (>6 months).

DETAILED DESCRIPTION:
This open-label clinical trial will compare outcomes of subjects with chronic stroke. Six subjects will be to treatment (n=3) groups. The treatment group will receive brain transplants of autologous ADSCs. Treatment group will receive rehabilitation after the transplantation. Subjects will be assessed by magnetic resonance imaging (MRI) and eight standardized stroke indices: National Institutes of Health Stroke Scale (NIHSS), ( Barthel Index )、 ( Berg balance scale )、 (Fugl - Meyer test )、(Action research arm test )、 (Purdue pegboard )、 ( grip strength measurement ) 、(somatosensory evoked potential, SSEP) at 1 month, 3 months, and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* stroke investigators with age 65 to 80 years
* history of stroke between six months and 10 years
* Systolic pressure and Diastolic pressure were maintained under 160 mmHg and 110 mmHg
* INR < 2.5, platelets counts 1-5 x 10^5/μl
* Damaged area range between 0.5 cm to 6 cm by brain MRI

Exclusion Criteria:

* Pregnant women
* Investigators with AIDS, cancer, liver dysfunction
* Others can't fit into the trial evaluate by investigator

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Neurological function | 6 months
  Blood biochemical, Neurobehavioral examination (NIH Stroke Scale 16-20)

CONTACTS AND LOCATIONS:
Overall Officials: Hualien T Hospital, Principal Investigator — Hualien Tzu Chi General Hospital
Locations (2):
- Taiwan (2):
  - Gwo Xi Stem Cell Applied Technology Co., Ltd., Hsinchu
  - Hualien Tzu Chi Hospital, Hualien City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiu TL, Baskaran R, Tsai ST, Huang CY, Chuang MH, Syu WS, Harn HJ, Lin YC, Chen CH, Huang PC, Wang YF, Chuang CH, Lin PC, Lin SZ. Intracerebral transplantation of autologous adipose-derived stem cells for chronic ischemic stroke: A phase I study. J Tissue Eng Regen Med. 2022 Jan;16(1):3-13. doi: 10.1002/term.3256. Epub 2021 Oct 21. PMID 34644444